CLINICAL TRIAL: NCT01851694
Title: Determination of Beta-cell Responsiveness to the Incretin Hormones GLP-1 and GIP in Cystic Fibrosis
Brief Title: Beta-cell Response to Incretin Hormones in Cystic Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Michael R. Rickels, MD, MS, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 817585
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis; Pancreatic Insufficiency
Keywords: Cystic Fibrosis; Diabetes; Pancreatic insufficiency; Cystic Fibrosis with Normal Glucose Tolerance; Non-Cystic Fibrosis control group
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Diabetes Mellitus | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 Incretin Hormone (Experimental): The incretin, Glucagon-Like-peptide-1 (GLP-1) will be infused into the veins starting 30 minutes prior to initiating the GPA test. This infusion will continue for a total of 90 mins. (during the GPA for 230 mg/dL glucose levels) and then this will be stopped. The GPA test will be performed for the 340 mg/dL glucose levels but no incretin will be infused during this part of the test. These data will be compared when the subject repeats the GPA test with a placebo (saline or salt containing solution) infusion.
  Interventions: Drug: GLP-1
- GIP Incretin Hormone (Experimental): The incretin, Glucose-dependent Insulinotropic Polypeptide (GIP) will be infused into the veins starting 30 minutes prior to initiating the GPA test. This infusion will continue for a total of 90 mins (during the GPA for 230 mg/dL glucose levels) and then this will be stopped. The GPA test will be performed for the 340 mg/dL glucose levels but no incretin will be infused during this part of the test. These data will be compared when the subject repeats the GPA test with a placebo (saline or salt containing solution) infusion.
  Interventions: Drug: GIP

INTERVENTIONS:
Drug: GLP-1 — Each subject in this arm will receive GLP-1 infusion and a placebo infusion during a GPA test.
  Arms: GLP-1 Incretin Hormone
Drug: GIP — Each subject in this arm will receive GIP infusion and placebo during a GPA test.
  Other Names: Glucose-dependent insulinotrophic polypeptide
  Arms: GIP Incretin Hormone

SUMMARY:
In recent years, diabetes has emerged as one of the most significant co-diseases that many Cystic Fibrosis (CF) patients develop. Type 1 (T1D) and Type 2 (T2D) diabetes results when either the body does not make enough insulin or the body does not respond correctly to this insulin, respectively. Insulin is a hormone which is made by cells in the pancreas and helps carry glucose (sugar) from the food we eat to the cells of the body for energy. While cystic fibrosis related diabetes (CFRD) has many features similar to both T1D and T2D, patients with CF may not have the same symptoms as either T1D or T2D patients. Currently, there is little understanding of CFRD and the best options for treatment remain unclear.

The purpose of this research study is to examine and understand the various mechanisms that contribute to CFRD and gain a better understanding of potential means to treat CFRD. In particular, we plan to study the effects of incretin hormones that can enhance insulin production in CF patients.

Enrollment is complete for the protocol as initially written. In order to further study the role of the incretin hormone on Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) function , we have received approval to extend our investigation to include the following study groups:

* Cystic Fibrosis participants with normal glucose tolerance
* Non-Cystic Fibrosis controls

DETAILED DESCRIPTION:
Previously, cystic fibrosis related diabetes (CFRD) was considered to be a consequence of damage to the pancreas therefore the cells contained in the pancreas--i.e.--islets that house beta cells, which make and release insulin (similar to T1D). Recent evidence suggests that other factors may also be associated that are similar to those with T2D. For example, patients with T2D, have decreased secretion of incretins, hormones released by the small intestine in response to nutrients from food which act, among other things, to increase insulin secretion from Beta cells of the pancreas. When patients with T2D are treated with incretin hormones, their pancreatic Beta cells release more insulin (measured as 'second phase insulin secretion'). Currently, we do not know if patients with CFRD have decreased incretin secretion like T2D or if treating CFRD patients with incretin hormones will improve their insulin levels. This study will measure insulin release from the Beta cells from CFRD patients (second phase insulin secretion) that are being given incretin hormones in the veins. This will be compared with insulin release when the same patients are given a placebo (salt containing solution). The patients and the research team will not know what is being given until all the results are collected. The results will provide unbiased evidence if incretins will help improve insulin release in CFRD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of cystic fibrosis, defined by positive sweat test or CFTR mutation analysis according to CFF diagnostic criteria,
2. Age greater than or equal to 18y on date of consent
3. Pancreatic insufficiency
4. Recent OGTT consistent with Indeterminate-GT, IGT, CFRD w/o fasting hyperglycemia, or an established diagnosis of CFRD without fasting hyperglycemia
5. For female subjects, negative urine pregnancy test at enrollment.

Control Subjects:

1. No history of cystic fibrosis.
2. Age ≥ 18y on date of consent.
3. Recent OGTT consistent with NGT.
4. For female subjects, negative urine pregnancy test at enrollment.

Exclusion Criteria:

1. Established diagnosis of non-CF diabetes (i.e. T1D) or CFRD with fasting hyperglycemia (fasting glucose greater than126 mg/dL)
2. History of clinically symptomatic pancreatitis within last year
3. Prior lung or liver transplant
4. Severe CF liver disease, as defined by portal hypertension
5. Fundoplication-related dumping syndrome
6. Medical co-morbidities that are not CF-related or are unstable per investigator opinion (i.e. history of bleeding disorders, immunodeficiency)
7. Acute illness or changes in therapy (including antibiotics) within 6 weeks prior to study procedures
8. Treatment with oral or intravenous corticosteroids within 6 weeks of study
9. Hemoglobin less than10g/dL, within 90 days of Visit 1 or at Screening
10. Abnormal renal function, within 90 days of Visit 1 or at Screening; defined as Creatinine greater than 2x upper limit of normal (ULN) or potassium greater than 5.5mEq/L on non-hemolyzed specimen
11. Inability to perform study specific procedures (MMTT, GPA)
12. Subjects, who in study team opinion, may be non-compliant with study procedures.

Control Subjects who will be exposed to GIP only:

1. History of clinically symptomatic pancreatitis.
2. History of liver disease.
3. History of any illness or condition that, in the opinion of the investigator might confound the results of the study or pose an additional risk to the subject.
4. Hemoglobin <10g/dL, within 90 days of GPA test or at Screening.
5. Abnormal renal function, within 90 days of GPA test or at Screening; defined as creatinine > 2x upper limit of normal (ULN) or potassium > 5.5mEq/L on non-hemolyzed specimen.
6. Inability to perform study specific procedures (MMTT, GPA).
7. subjects, who in study team opinion, may be non-compliant with study procedures.
8. elevation of serum amylase or lipase > 1.5x ULN within 90 days of GPA test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-05; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Second-phase insulin response during GPA test | 5 hours
  The key endpoint of interest will be the change in second phase insulin response derived from the Glucose-Potentiated Arginine (GPA) test. The GPA test will measure insulin (and other glucose controlling hormones) which will be a measure of pancreatic endocrine function in response to injection of arginine. Arginine is a naturally occurring amino acid (substance) in the body. It will be given in the veins to make the pancreas secrete insulin. After the first injection of arginine, a glucose infusion will be started in order to raise the level of sugar in the blood to 230 mg/dl. Once the level is achieved, arginine will be injected again and blood samples are measured. After a 2 hour break, the glucose infusion will be started to achieve a blood sugar of 340mg/dl and arginine injection will be repeated. Comparison of responses with incretin vs. placebo will be performed using statistical methods, specifically, paired t-test or Wilcoxon matched pair test.

SECONDARY OUTCOMES:
Change in insulin secretion among CF groups | 5 hours
  The change in second phase insulin secretion induced by incretins will be compared among the different subgroups of patients with CF (Ind-GT, IGT, and early CFRD) groups using nonparametric comparison of changes in slope, estimated using Mann-Whitney methods.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Rickels, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- Children's Hospital of Philadelphia and University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of enrollment, once our data has been analyzed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon completion of enrollment, once our data has been analyzed. Informed Consent has already been shared.
Access Criteria: Will upload on clinical trials.gov and attach to results section. Informed Consent has already been shared on ct.gov.

REFERENCES:
- [Derived] Nyirjesy SC, Peleckis AJ, Eiel JN, Gallagher K, Doliba A, Tami A, Flatt AJ, De Leon DD, Hadjiliadis D, Sheikh S, Stefanovski D, Gallop R, D'Alessio DA, Rubenstein RC, Kelly A, Rickels MR. Effects of GLP-1 and GIP on Islet Function in Glucose-Intolerant, Pancreatic-Insufficient Cystic Fibrosis. Diabetes. 2022 Oct 1;71(10):2153-2165. doi: 10.2337/db22-0399. PMID 35796669

DOCUMENTS (1):
  • Informed Consent Form (2018-12-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT01851694/ICF_000.pdf